CLINICAL TRIAL: NCT00408421
Title: Duloxetine 60 to 120 mg Versus Placebo in the Treatment of Patients With Osteoarthritis Knee Pain
Brief Title: Duloxetine Versus Placebo for Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10546; F1J-MC-HMEP
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis Knee Pain
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): duloxetine 30 mg, daily (QD), by mouth (PO) for 1 week then duloxetine 60 mg QD, PO for 6 weeks then duloxetine 60 mg or 120 mg QD, PO for 6 weeks
  Interventions: Drug: Duloxetine
- B (Placebo Comparator): placebo daily (QD), by mouth (PO) for 13 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Duloxetine
  Other Names: LY248686; Cymbalta
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
The primary purpose of this study is to determine if duloxetine reduces pain severity in patients with osteoarthritis knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients with osteoarthritis knee pain.

Exclusion Criteria:

* Cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
* Acute liver injury (such as hepatitis) or severe cirrhosis.
* Previous exposure to duloxetine.
* Body Mass Index (BMI) over 40.
* Major depressive disorder.
* Daily use of narcotics.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chandler, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Walnut Creek, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuart, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morton Grove, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billerica, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waltham, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westborough, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edison, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stratford, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waco, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita Falls, Texas
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași

REFERENCES:
- [Derived] Yue L, Wang J, Enomoto H, Fujikoshi S, Alev L, Cheng YY, Skljarevski V. The Clinical Relevance of Pain Severity Changes: Is There Any Difference Between Asian and Caucasian Patients With Osteoarthritis Pain? Pain Pract. 2020 Feb;20(2):129-137. doi: 10.1111/papr.12835. Epub 2019 Nov 20. PMID 31505082
- [Derived] Williamson OD, Schroer M, Ruff DD, Ahl J, Margherita A, Sagman D, Wohlreich MM. Onset of response with duloxetine treatment in patients with osteoarthritis knee pain and chronic low back pain: a post hoc analysis of placebo-controlled trials. Clin Ther. 2014 Apr 1;36(4):544-51. doi: 10.1016/j.clinthera.2014.02.009. Epub 2014 Mar 17. PMID 24650448
- [Derived] Hochberg MC, Wohlreich M, Gaynor P, Hanna S, Risser R. Clinically relevant outcomes based on analysis of pooled data from 2 trials of duloxetine in patients with knee osteoarthritis. J Rheumatol. 2012 Feb;39(2):352-8. doi: 10.3899/jrheum.110307. Epub 2011 Dec 1. PMID 22133624
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo daily (QD), by mouth (PO) for 13 weeks
- Duloxetine 60 mg: Patients randomly assigned to duloxetine 60 mg daily (QD) started on duloxetine 30 mg QD for 1 week and then titrated up to duloxetine 60 mg QD for the following 6 weeks of the treatment phase. Beginning at Week 7, patients on duloxetine 60 mg QD were re-randomized to either duloxetine 60 mg QD or duloxetine 120 mg QD.
- Duloxetine 120 mg: Beginning at Week 7, patients receiving duloxetine 60 mg daily (QD) were re-randomized to either duloxetine 60 mg QD or duloxetine 120 mg QD
Period: Treatment Initial Randomization
Arm/Group | Placebo | Duloxetine 60 mg | Duloxetine 120 mg
Started | 120 | 111 | 0
Completed | 103 (Pre-Re-Randomization (Visit 4)) | 89 (Pre-Re-Randomization (Visit 4)) | 0 (Patients weren't randomized to Duloxetine 120 mg until Visit 4.)
Not Completed | 17 | 22 | 0
Not completed — Adverse Event | 5 | 9 | 0
Not completed — Lack of Efficacy | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 0
Not completed — Entry Criteria Not Met | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0
Period: Treatment Re-Randomization
Arm/Group | Placebo | Duloxetine 60 mg | Duloxetine 120 mg
Started | 103 | 46 | 43
Completed | 96 | 39 | 38
Not Completed | 7 | 7 | 5
Not completed — Adverse Event | 2 | 2 | 4
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 3 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine 60mg /120mg: Patients randomly assigned to duloxetine 60 mg QD started on duloxetine 30 mg QD for 1 week and then titrated up to duloxetine 60 mg QD for the following 6 weeks of the treatment phase. Beginning Week 7, patients assigned to duloxetine 60 mg were re-randomized to receive either duloxetine 60 mg or duloxetine 120 mg, and when combined are considered the Duloxetine 60mg/120mg group.
- Total: Total of all reporting groups
Arm/Group | Placebo | Duloxetine 60mg /120mg | Total
Number analyzed (Participants) | 120 | 111 | 231
Age Continuous [Mean (Standard Deviation); unit: years] | 62.48 (9.30) | 62.07 (9.63) | 62.28 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 70 | 151
  Male | 39 | 41 | 80
Race/Ethnicity, Customized [Number; unit: participants]
  African | 6 | 6 | 12
  Caucasian | 100 | 94 | 194
  East Asian | 3 | 0 | 3
  Hispanic | 10 | 9 | 19
  Native American | 1 | 2 | 3
Non Steroidal Anti Inflammatory Drug Use [Number; unit: participants]
  Yes | 59 | 58 | 117
  No | 61 | 53 | 114
Brief Pain Inventory (BPI) Average Pain [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). The Average Pain Score reflects the average pain score over the last 24-hours.
  units on a scale | 6.23 (1.54) | 6.16 (1.58) | 6.20 (1.56)
Duration of Osteoarthritis (OA) Pain Since Onset [Mean (Standard Deviation); unit: years] | 9.30 (8.27) | 9.04 (8.72) | 9.17 (8.47)
Duration of Osteoarthritis Since Diagnosis [Mean (Standard Deviation); unit: years] | 7.09 (7.20) | 6.94 (8.38) | 7.01 (7.77)
Height [Mean (Standard Deviation); unit: centimeters] | 164.67 (9.49) | 167.01 (8.81) | 165.79 (9.22)
Patient Global Impressions of Severity (PGI-Severity) [Mean (Standard Deviation); unit: units on a scale] — Measures patient's perception of severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (extremely ill).
  units on a scale | 2.40 (1.64) | 2.21 (1.51) | 2.31 (1.58)
Weekly Mean of 24-Hour Average Pain Severity [Mean (Standard Deviation); unit: units on a scale] — This is an ordinal scale assessing the 24-hour average pain with scores from 0 (no pain) to 10 (worst possible pain).
  units on a scale | 6.18 (1.32) | 6.10 (1.34) | 6.14 (1.33)
Weight [Mean (Standard Deviation); unit: kilograms] | 85.66 (15.12) | 85.57 (16.17) | 85.61 (15.60)

OUTCOME MEASURES:

1. Primary Outcome: Weekly Change From Baseline in the 24-Hour Average Pain Rating Using an 11-Point Numerical Likert Scale Patient Diary
Description: This is an ordinal scale assessing the 24-hour average pain with scores from 0 (no pain) to 10 (worst possible pain).
Time Frame: Over 13 Weeks
Population: Analyses were conducted on an intent-to-treat basis. All randomized patients with a baseline and at least one non-missing post-baseline value for the specific outcome measure were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 119 | 103
units on a scale
  Week 1 (Change from Baseline): N=119, N=103 | -0.36 (0.15) | -0.84 (0.16)
  Week 2 (Change from Baseline): N=112, N=101 | -0.95 (0.15) | -1.54 (0.16)
  Week 3 (Change from Baseline): N=110, N=97 | -1.23 (0.15) | -1.85 (0.16)
  Week 4 (Change from Baseline): N=109, N=96 | -1.42 (0.15) | -2.10 (0.16)
  Week 5 (Change from Baseline): N=107, N=90 | -1.55 (0.15) | -2.29 (0.16)
  Week 6 (Change from Baseline): N=108, N=92 | -1.61 (0.15) | -2.41 (0.16)
  Week 7 (Change from Baseline): N=107, N=92 | -1.72 (0.15) | -2.60 (0.16)
  Week 8 (Change from Baseline): N=86, N=78 | -1.93 (0.15) | -2.60 (0.16)
  Week 9 (Change from Baseline): N=98, N=81 | -1.89 (0.15) | -2.73 (0.17)
  Week 10 (Change from Baseline): N=99, N=80 | -1.94 (0.16) | -2.74 (0.17)
  Week 11 (Change from Baseline): N=99, N=81 | -1.94 (0.16) | -2.89 (0.17)
  Week 12 (Change from Baseline): N=98, N=80 | -1.98 (0.16) | -2.93 (0.17)
  Week 13 (Change from Baseline): N=97, N=75 | -2.08 (0.16) | -2.92 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; Null hypothesis: the difference in 24-hour average pain score between duloxetine and placebo treatment groups at last visit of treatment phase is zero. This study will have at least 80% power to detect a treatment group difference of 1.0 point in the baseline-to-endpoint mean change on the weekly mean of 24-hour average pain severity between duloxetine and placebo treatment groups based on Baseline Observation Carried Forward (BOCF); Test type: Superiority or Other; p < 0.001, Mixed-Effects Model Repeated Measures — P-value for treatment effect at last visit. Effects evaluated based on 2-sided significance level=0.05. Model: treatment, NSAID use, investigator, week, treatment-by-week interaction, baseline score and baseline-by-week interaction; No adjustments for multiple comparisons were made

2. Secondary Outcome: Patient Global Impression of Improvement at 13 Week Endpoint
Description: A scale that measures the patient's perception of improvement at the time of assessment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: 13 Weeks
Population: Analysis was conducted on an intent-to-treat basis. Missing data were imputed using a Last Observation Carried Forward approach. All randomized patients with a baseline and at least one non-missing post-baseline value for the specific for the specific outcome measure were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 114 | 104
units on a scale | 2.91 (0.12) | 2.38 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; An analysis of covariance (ANCOVA) model was used which contains the terms of treatment, NSAID use (Yes/No), PGI severity at baseline, and investigator. Type III sum-of-squares for the least-squares mean (LSMean) was used to test the null hypothesis that there is no treatment difference on the mean outcome measure at endpoint; Test type: Superiority or Other; p = 0.001, ANCOVA — Treatment effects and interaction effects were evaluated based on a two-sided significance level of 0.05. No adjustments for multiple comparisons were made; Mean Difference (Net) = -0.53, 95% CI [-0.84 to -0.21]

3. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Pain Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the patient. The pain subscale has 5 questions on pain associated with every day tasks. Each question is answered using a 5-point Likert scale (0 to 4). The pain subscale has a range of scores of 0 (none) to 20 (extreme).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
units on a scale
  Baseline | 10.95 (3.00) | 10.98 (3.33)
  Change from Baseline | -3.19 (3.87) | -4.62 (4.34)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; An analysis of covariance (ANCOVA) model was used which contains the terms of treatment, NSAID use (Yes/No), the outcome score at baseline, and investigator. Type III sum-of-squares for the least-squares mean (LSMean) was used to test the null hypothesis that there is no treatment difference on the mean change from baseline to the endpoint of the outcome measure; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Change from Baseline. Treatment effects and interaction effects were evaluated based on a two-sided significance level of 0.05. No adjustments for multiple comparisons were made. Change=Endpoint-Baseline; Mean Difference (Net) = -1.41, 95% CI [-2.33 to -0.48] — Mean Difference = Duloxetine minus Placebo

4. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Stiffness Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the patient. The stiffness subscale has 2 questions on stiffness associated with time of day (morning versus later in the day). Each question is answered using a 5-point Likert scale (0 to 4). The pain subscale has a range of scores of 0 (none) to 8 (extreme).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 107
units on a scale
  Baseline | 4.80 (1.62) | 4.74 (1.59)
  Change from Baseline | -1.37 (1.88) | -1.97 (2.16)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.65, 95% CI [-1.09 to -0.22] — Mean Difference = Duloxetine minus Placebo

5. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Physical Function Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the patient. The physical function subscale has 17 questions on physical function difficulties with every day tasks. Each question is answered using a 5-point Likert scale (0 to 4). The physical function subscale has a range of scores of 0 (none) to 68 (extreme).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 115 | 104
units on a scale
  Baseline | 38.50 (10.12) | 39.10 (11.06)
  Change from Baseline | -11.58 (12.39) | -16.46 (14.65)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -5.18, 95% CI [-8.33 to -2.03] — Mean Difference = Duloxetine minus Placebo

6. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Total Score
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the patient. The index has 24 questions. Each question is answered using a 5-point Likert scale (0 to 4). The Total score has a range from 0 (none) to 96 (extreme).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 107
units on a scale
  Baseline | 53.36 (14.73) | 53.72 (16.51)
  Change from Baseline | -15.93 (17.53) | -22.19 (20.78)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -6.42, 95% CI [-10.72 to -2.11] — Mean Difference = Duloxetine minus Placebo

7. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Weekly Mean of the 24-Hour Worst Pain Score
Description: This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). The value is the change from baseline in the weekly mean of the 24-hour worst pain score on the scale.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 119 | 108
units on a scale
  Baseline | 7.54 (1.32) | 7.45 (1.12)
  Change from Baseline | -2.01 (2.02) | -2.81 (2.40)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.83, 95% CI [-1.40 to -0.25] — Mean Difference = Duloxetine minus Placebo

8. Secondary Outcome: Weekly Change From Baseline in the 24-Hour Worst Pain Score
Description: as for outcome 7
Time Frame: Over 13 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 119 | 103
units on a scale
  Week 1 (Change from Baseline): N=119, N=103 | -0.31 (0.16) | -0.82 (0.17)
  Week 2 (Change from Baseline): N=112, N=101 | -0.92 (0.16) | -1.57 (0.17)
  Week 3 (Change from Baseline): N=110, N=97 | -1.20 (0.17) | -1.99 (0.17)
  Week 4 (Change from Baseline): N=109, N=96 | -1.41 (0.17) | -2.26 (0.17)
  Week 5 (Change from Baseline): N=107, N=90 | -1.49 (0.17) | -2.40 (0.18)
  Week 6 (Change from Baseline): N=108, N=92 | -1.57 (0.17) | -2.58 (0.18)
  Week 7 (Change from Baseline): N=107, N=92 | -1.71 (0.17) | -2.82 (0.18)
  Week 8 (Change from Baseline): N=86, N=78 | -1.95 (0.17) | -2.82 (0.18)
  Week 9 (Change from Baseline): N=98, N=81 | -1.90 (0.17) | -2.94 (0.18)
  Week 10 (Change from Baseline): N=99, N=80 | -1.97 (0.17) | -3.00 (0.19)
  Week 11 (Change from Baseline): N=99, N=81 | -2.03 (0.17) | -3.12 (0.19)
  Week 12 (Change from Baseline): N=98, N=80 | -2.04 (0.17) | -3.14 (0.19)
  Week 13 (Change from Baseline): N=97, N=75 | -2.18 (0.18) | -3.19 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; Test type: Superiority or Other; p < 0.001, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; No adjustments for multiple comparisons were made

9. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Weekly Mean of 24-Hour Average Pain in the Re-Randomized Treatment Phase
Description: This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). This value is the change from baseline in the weekly mean of the 24-hour average pain score on the scale.
Time Frame: Baseline and 13 Weeks
Population: Analysis was conducted on an intent-to-treat basis in the re-randomized patients. Missing data were imputed using a Last Observation Carried Forward approach. All randomized patients with a baseline and at least one non-missing post-baseline value for the specific for the specific outcome measure were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 2 - Duloxetine 60mg | Group 3 - Duloxetine 120mg
Number analyzed (Participants) | 46 | 43
units on a scale
  Baseline | 5.96 (1.41) | 6.22 (1.37)
  Change from Baseline | -2.46 (1.99) | -3.44 (1.76)
Statistical Analysis 1: Comparison: Group 2 - Duloxetine 60mg vs Group 3 - Duloxetine 120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.039, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.87, 95% CI [-1.69 to -0.05] — Mean Difference = Duloxetine minus Placebo

10. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Clinical Global Impression of Severity
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 103
units on a scale
  Baseline | 2.62 (1.47) | 2.71 (1.56)
  Change from Baseline | -0.21 (1.28) | -0.70 (1.30)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.35, 95% CI [-0.56 to -0.14] — Mean Difference = Duloxetine minus Placebo

11. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory (BPI) - Worst Pain Score
Description: A self-reported scale that measures the severity of pain based on the worst pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
units on a scale
  Baseline | 7.64 (1.45) | 7.60 (1.38)
  Change from Baseline | -2.15 (2.17) | -3.17 (2.72)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -1.06, 95% CI [-1.66 to -0.46] — Mean Difference = Duloxetine minus Placebo

12. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory - Least Pain Score
Description: A self-reported scale that measures the severity of pain based on the least pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
units on a scale
  Baseline | 5.09 (2.00) | 5.07 (2.12)
  Change from Baseline | -1.60 (2.13) | -2.30 (2.50)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.76, 95% CI [-1.28 to -0.24] — Mean Difference = Duloxetine minus Placebo

13. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory - Average Pain Score
Description: A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 116 | 107
units on a scale
  Baseline | 6.25 (1.55) | 6.19 (1.59)
  Change from Baseline | -1.77 (2.19) | -2.71 (2.43)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.97, 95% CI [-1.52 to -0.42] — Mean Difference = Duloxetine minus Placebo

14. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory - Pain Right Now Score
Description: A self-reported scale that measures the severity of pain based on the pain right now. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
units on a scale
  Baseline | 6.02 (2.17) | 5.77 (2.14)
  Change from Baseline | -2.26 (2.83) | -2.94 (2.55)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.91, 95% CI [-1.50 to -0.32] — Mean Difference = Duloxetine minus Placebo

15. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference Score - General Activity
Description: A self-reported scale that measures the interference of pain in the past 24 hours on general acitivity. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 5.55 (2.23) | 5.50 (2.43)
  Change from Baseline | -1.97 (2.72) | -2.63 (2.50)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.019, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.71, 95% CI [-1.30 to -0.12] — Mean Difference = Duloxetine minus Placebo

16. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference Score - Mood
Description: A self-reported scale that measures the interference of pain in the past 24 hours on mood. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 4.22 (2.74) | 4.06 (2.66)
  Change from Baseline | -1.69 (2.66) | -1.95 (2.54)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.164, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.40, 95% CI [-0.97 to 0.17] — Mean Difference = Duloxetine minus Placebo

17. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference Score - Walking Ability
Description: A self-reported scale that measures the interference of pain in the past 24 hours on walking ability. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 6.00 (2.29) | 5.72 (2.26)
  Change from Baseline | -2.36 (2.73) | -2.80 (2.87)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.049, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.63, 95% CI [-1.25 to 0.00] — Mean Difference = Duloxetine minus Placebo

18. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference Score - Normal Work
Description: A self-reported scale that measures the interference of pain in the past 24 hours on normal work. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 5.80 (2.08) | 5.63 (2.32)
  Change from Baseline | -2.25 (2.48) | -2.66 (2.56)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.093, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.51, 95% CI [-1.10 to 0.08] — Mean Difference = Duloxetine minus Placebo

19. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference Score - Relations With Other People
Description: A self-reported scale that measures the interference of pain in the past 24 hours on relations with other people. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 3.27 (2.82) | 3.05 (2.81)
  Change from Baseline | -1.30 (2.48) | -1.43 (2.51)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.287, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.29, 95% CI [-0.82 to 0.24] — Mean Difference = Duloxetine minus Placebo

20. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference Score - Sleep
Description: A self-reported scale that measures the interference of pain in the past 24 hours on sleep. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 4.16 (2.98) | 4.23 (2.91)
  Change from Baseline | -1.57 (2.87) | -2.18 (2.95)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.033, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.64, 95% CI [-1.23 to -0.05] — Mean Difference = Duloxetine minus Placebo

21. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference Score - Enjoyment of Life
Description: A self-reported scale that measures the interference of pain in the past 24 hours on enjoyment of life. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 4.04 (2.89) | 4.42 (3.06)
  Change from Baseline | -1.39 (2.89) | -2.38 (3.03)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.78, 95% CI [-1.40 to -0.15] — Mean Difference = Duloxetine minus Placebo

22. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Average Interference
Description: A self-reported scale that measures interference of pain on average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The average Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 104
units on a scale
  Baseline | 4.72 (2.08) | 4.66 (2.16)
  Change from Baseline | -1.79 (2.10) | -2.29 (2.18)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.029, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.56, 95% CI [-1.06 to -0.06] — Mean Difference = Duloxetine minus Placebo

23. Secondary Outcome: Response to Treatment - The Number of Participants With a >= 30% Reduction of Weekly Mean in 24-Hour Average Pain Severity Ratings
Description: Number of participants who experienced a response to treatment, which was defined as having a >=30% reduction of the weekly mean in 24-hour average pain severity ratings. This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain).
Time Frame: Over 13 Weeks
Population: as for outcome 2
Measure: Number; unit: participants who responded
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 119 | 108
participants who responded | 53 | 64
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; This study will also have at least 85% power to detect a treatment group difference of 25% in the response rates (≥30% reduction from baseline) based on the weekly mean of 24-hour average pain severity between duloxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.033, Fisher Exact

24. Secondary Outcome: Response to Treatment - The Number of Participants With a >=30% Reduction of Weekly Mean in 24-Hour Average Pain Severity Ratings in the Re-Randomized Treatment Phase
Description: Number of participants who experienced a response to treatment, which was defined as having a >=30% reduction of the weekly mean in 24-hour average pain severity ratings. Response to treatment over the last 6 weeks of the trial (after patients were re-randomized) were compared to baseline measures.
Time Frame: Over 13 Weeks
Population: Number of re-randomized patients with non-missing response values.
Measure: Number; unit: participants who responded
Arm/Group | Group 2 - Duloxetine 60mg | Group 3 - Duloxetine 120mg
Number analyzed (Participants) | 45 | 42
participants who responded | 26 | 32
Statistical Analysis 1: Comparison: Group 2 - Duloxetine 60mg vs Group 3 - Duloxetine 120mg; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.075, Fisher Exact

25. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Medical Outcomes Study Short Form-36 (SF-36) - Mental Health Component Summary
Description: A self-reported questionnaire that consists of 36 questions covering 8 health domains. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. The mental component summary (MCS) has been constructed based on the 8 SF-36 domains.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 113 | 103
units on a scale
  Baseline | 56.58 (10.38) | 56.43 (10.36)
  Change from Baseline | -1.03 (9.34) | 1.06 (8.84)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.088, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 1.83, 95% CI [-0.28 to 3.94] — Mean Difference = Duloxetine minus Placebo

26. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Medical Outcomes Study Short Form-36 (SF-36) - Physical Component Summary
Description: A self-reported questionnaire that consists of 36 questions covering 8 health domains. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. The physical component summary (PCS) has been constructed based on the 8 SF-36 domains.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 113 | 103
units on a scale
  Baseline | 30.57 (8.13) | 31.56 (8.90)
  Change from Baseline | 6.36 (9.24) | 7.71 (8.61)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.080, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 1.87, 95% CI [-0.22 to 3.96] — Mean Difference = Duloxetine minus Placebo

27. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Euro-Quality of Life - 5 Dimensions (EQ-5D): US Based Index Score
Description: The EQ-5D is an assessment of one's overall health. Consists of 5 items. Patients choose 1 of 3 options that best describe the status of each item. The EQ-5D US based index scores range from -0.11 to 1.0 where a score of 1.0 indicates perfect health. A positive change from baseline indicates health improvement.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 114 | 103
units on a scale
  Baseline | 0.70 (0.16) | 0.68 (0.18)
  Change from Baseline | 0.07 (0.16) | 0.14 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 0.06, 95% CI [0.03 to 0.10] — Mean Difference = Duloxetine minus Placebo

28. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Beck Depression Inventory-II - Total Score
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 107
units on a scale
  Baseline | 5.64 (5.89) | 5.49 (6.84)
  Change from Baseline | -0.97 (4.34) | -1.26 (3.88)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.641, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.23, 95% CI [-1.19 to 0.74] — Mean Difference = Duloxetine minus Placebo

29. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale
Description: A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 112 | 101
units on a scale
  Baseline | 5.36 (3.86) | 4.59 (4.02)
  Change from Baseline | -0.93 (2.58) | -1.15 (3.12)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.193, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.47, 95% CI [-1.17 to 0.24] — Mean Difference = Duloxetine minus Placebo

30. Secondary Outcome: Statistically Significant Change From Baseline to 13 Week Endpoint in Laboratory Data - Chemistry Analytes: Alkaline Phosphatase
Description: Change from baseline to endpoint in alkaline phosphatase using central laboratory reference ranges.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/Liter
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
Units/Liter
  Baseline | 76.97 (21.75) | 78.59 (20.83)
  Change from Baseline | -1.94 (10.54) | 2.08 (12.95)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; An analysis of variance (ANOVA) model was used which contains the terms of treatment and investigator. Rank-transformed data will be used in the analysis given the view that the change scores for most of the laboratory analytes are not normally distributed. Type III sum-of-squares for the least-squares mean (LSMean) was used to test the null hypothesis that there is no treatment difference on the mean change from baseline to the endpoint of the outcome measure; Test type: Superiority or Other; p = 0.003, ANOVA — [p-value comment as in outcome 3, analysis 1]; ANOVA on ranked data

31. Secondary Outcome: Statistically Significant Change From Baseline to 13 Week Endpoint in Laboratory Data - Chemistry Analytes: Uric Acid
Description: Change from baseline to endpoint in uric acid using central laboratory reference ranges.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
micromole/Liter
  Baseline | 314.57 (77.12) | 322.77 (95.86)
  Change from Baseline | 6.82 (48.99) | -5.00 (47.90)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 30, analysis 1]; Test type: Superiority or Other; p = 0.026, ANOVA — [p-value comment as in outcome 3, analysis 1]; ANOVA on ranked data

32. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Vital Signs - Pulse Rate
Description: Pulse rate (heart rate) measured in the sitting position.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
beats per minute
  Baseline | 70.07 (8.32) | 69.75 (8.33)
  Change from Baseline | 1.26 (7.52) | 2.02 (8.48)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; An analysis of variance (ANOVA) model was used which contains the terms of treatment and investigator. Type III sum-of-squares for the least-squares mean (LSMean) was used to test the null hypothesis that there is no treatment difference on the mean change from baseline to the endpoint of the outcome measure; Test type: Superiority or Other; p = 0.459, ANOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 0.80, 95% CI [-1.32 to 2.92] — Mean Difference = Duloxetine minus Placebo

33. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Vital Signs - Blood Pressure (BP) Diastolic
Description: Diastolic blood pressure measured in the sitting position.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
mm Hg
  Baseline | 76.44 (9.78) | 77.00 (8.82)
  Change from Baseline | -0.38 (8.73) | 0.95 (8.46)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 32, analysis 1]; Test type: Superiority or Other; p = 0.326, ANOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 1.09, 95% CI [-1.10 to 3.28] — Mean Difference = Duloxetine minus Placebo

34. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Vital Signs - Blood Pressure (BP) Systolic
Description: Systolic blood pressure measured in the sitting position.
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 117 | 107
mm Hg
  Baseline | 129.42 (14.44) | 128.27 (14.39)
  Change from Baseline | -2.29 (12.35) | 1.04 (14.02)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 32, analysis 1]; Test type: Superiority or Other; p = 0.069, ANOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 3.16, 95% CI [-0.25 to 6.56] — Mean Difference = Duloxetine minus Placebo

35. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Vital Signs - Weight
Time Frame: Baseline and 13 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo | Duloxetine 60mg /120mg
Number analyzed (Participants) | 118 | 107
kilograms
  Baseline | 85.56 (15.14) | 85.39 (16.25)
  Change from Baseline | -0.33 (2.24) | -0.79 (2.70)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 60mg /120mg; [analysis description as in outcome 32, analysis 1]; Test type: Superiority or Other; p = 0.107, ANOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.54, 95% CI [-1.20 to 0.12] — Mean Difference = Duloxetine minus Placebo

ADVERSE EVENTS:
Groups:
- Placebo: Placebo
- Duloxetine 60/120 mg QD: Duloxetine 60/120 mg QD
Arm/Group | Placebo | Duloxetine 60/120 mg QD
Serious Adverse Events (participants affected / at risk) | 2 | 1
Other Adverse Events (participants affected / at risk) | 49 | 55
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Duloxetine 60/120 mg QD
Myocardial infarction (Cardiac disorders) | 1/120 (1) | 0/111 (0)
Bronchitis (Infections and infestations) | 0/120 (0) | 1/111 (1)
Dehydration (Metabolism and nutrition disorders) | 1/120 (1) | 0/111 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/120 (0) | 1/111 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0/120 (0) | 1/111 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Duloxetine 60/120 mg QD
Lymphadenopathy (Blood and lymphatic system disorders) | 0/120 (0) | 1/111 (1)
Coronary artery disease (Cardiac disorders) | 1/120 (1) | 0/111 (0)
Palpitations (Cardiac disorders) | 1/120 (1) | 0/111 (0)
Ear pain (Ear and labyrinth disorders) | 1/120 (1) | 0/111 (0)
Hyperthyroidism (Endocrine disorders) | 1/120 (1) | 0/111 (0)
Vision blurred (Eye disorders) | 0/120 (0) | 2/111 (2)
Abdominal pain (Gastrointestinal disorders) | 2/120 (2) | 1/111 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0/120 (0) | 1/111 (1)
Constipation (Gastrointestinal disorders) | 0/120 (0) | 4/111 (4)
Diarrhoea (Gastrointestinal disorders) | 3/120 (3) | 5/111 (7)
Dry mouth (Gastrointestinal disorders) | 2/120 (2) | 2/111 (2)
Dyspepsia (Gastrointestinal disorders) | 1/120 (1) | 1/111 (1)
Flatulence (Gastrointestinal disorders) | 0/120 (0) | 2/111 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/120 (1) | 1/111 (1)
Haemorrhoids (Gastrointestinal disorders) | 0/120 (0) | 1/111 (1)
Hiatus hernia (Gastrointestinal disorders) | 0/120 (0) | 1/111 (1)
Nausea (Gastrointestinal disorders) | 2/120 (2) | 7/111 (7)
Stomatitis (Gastrointestinal disorders) | 1/120 (1) | 1/111 (1)
Toothache (Gastrointestinal disorders) | 1/120 (1) | 0/111 (0)
Asthenia (General disorders) | 0/120 (0) | 2/111 (3)
Chest pain (General disorders) | 1/120 (1) | 0/111 (0)
Chills (General disorders) | 0/120 (0) | 1/111 (1)
Condition aggravated (General disorders) | 0/120 (0) | 1/111 (1)
Fatigue (General disorders) | 1/120 (1) | 7/111 (8)
Oedema peripheral (General disorders) | 1/120 (1) | 2/111 (2)
Pain (General disorders) | 1/120 (1) | 0/111 (0)
Pyrexia (General disorders) | 0/120 (0) | 1/111 (1)
Swelling (General disorders) | 1/120 (1) | 0/111 (0)
Biliary colic (Hepatobiliary disorders) | 1/120 (1) | 0/111 (0)
Hypersensitivity (Immune system disorders) | 1/120 (1) | 0/111 (0)
Seasonal allergy (Immune system disorders) | 0/120 (0) | 1/111 (1)
Bronchitis (Infections and infestations) | 2/120 (2) | 0/111 (0)
Cellulitis (Infections and infestations) | 1/120 (1) | 0/111 (0)
Fungal infection (Infections and infestations) | 1/120 (1) | 0/111 (0)
Influenza (Infections and infestations) | 1/120 (1) | 1/111 (1)
Molluscum contagiosum (Infections and infestations) | 1/120 (1) | 0/111 (0)
Nasopharyngitis (Infections and infestations) | 0/120 (0) | 1/111 (1)
Oral herpes (Infections and infestations) | 0/120 (0) | 1/111 (1)
Upper respiratory tract infection (Infections and infestations) | 2/120 (2) | 1/111 (1)
Viral infection (Infections and infestations) | 2/120 (2) | 0/111 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1/120 (1) | 0/111 (0)
Contusion (Injury, poisoning and procedural complications) | 0/120 (0) | 1/111 (1)
Fall (Injury, poisoning and procedural complications) | 1/120 (2) | 1/111 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1/120 (1) | 1/111 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1/120 (1) | 0/111 (0)
Blood creatine phosphokinase increased (Investigations) | 1/120 (1) | 2/111 (2)
Blood creatinine increased (Investigations) | 1/120 (1) | 0/111 (0)
Blood phosphorus decreased (Investigations) | 1/120 (1) | 0/111 (0)
Blood pressure increased (Investigations) | 0/120 (0) | 1/111 (1)
Blood uric acid increased (Investigations) | 1/120 (1) | 1/111 (1)
Liver function test abnormal (Investigations) | 0/120 (0) | 1/111 (1)
Weight decreased (Investigations) | 1/120 (1) | 0/111 (0)
Anorexia (Metabolism and nutrition disorders) | 0/120 (0) | 1/111 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1/120 (1) | 3/111 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 0/120 (0) | 1/111 (1)
Fluid retention (Metabolism and nutrition disorders) | 0/120 (0) | 1/111 (1)
Gout (Metabolism and nutrition disorders) | 0/120 (0) | 1/111 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0/120 (0) | 1/111 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0/120 (0) | 1/111 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0/120 (0) | 1/111 (1)
Increased appetite (Metabolism and nutrition disorders) | 2/120 (2) | 0/111 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/120 (3) | 1/111 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0/120 (0) | 1/111 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2/120 (2) | 0/111 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2/120 (2) | 1/111 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0/120 (0) | 1/111 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 1/111 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/120 (0) | 1/111 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0/120 (0) | 1/111 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1/120 (1) | 0/111 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1/120 (3) | 0/111 (0)
Diabetic neuropathy (Nervous system disorders) | 1/120 (1) | 0/111 (0)
Disturbance in attention (Nervous system disorders) | 0/120 (0) | 1/111 (1)
Dizziness (Nervous system disorders) | 2/120 (3) | 4/111 (4)
Headache (Nervous system disorders) | 1/120 (1) | 3/111 (3)
Hypersomnia (Nervous system disorders) | 0/120 (0) | 1/111 (1)
Hypoaesthesia (Nervous system disorders) | 2/120 (2) | 0/111 (0)
Judgement impaired (Nervous system disorders) | 0/120 (0) | 1/111 (1)
Lethargy (Nervous system disorders) | 1/120 (1) | 1/111 (2)
Memory impairment (Nervous system disorders) | 0/120 (0) | 1/111 (1)
Migraine (Nervous system disorders) | 2/120 (2) | 1/111 (1)
Nerve compression (Nervous system disorders) | 0/120 (0) | 1/111 (1)
Paraesthesia (Nervous system disorders) | 0/120 (0) | 1/111 (1)
Poor quality sleep (Nervous system disorders) | 0/120 (0) | 1/111 (1)
Sciatica (Nervous system disorders) | 1/120 (1) | 1/111 (1)
Serotonin syndrome (Nervous system disorders) | 1/120 (1) | 0/111 (0)
Sinus headache (Nervous system disorders) | 1/120 (2) | 0/111 (0)
Somnolence (Nervous system disorders) | 1/120 (1) | 5/111 (5)
Agitation (Psychiatric disorders) | 0/120 (0) | 1/111 (1)
Anxiety (Psychiatric disorders) | 0/120 (0) | 1/111 (1)
Apathy (Psychiatric disorders) | 0/120 (0) | 1/111 (1)
Depression (Psychiatric disorders) | 1/120 (2) | 0/111 (0)
Disorientation (Psychiatric disorders) | 0/120 (0) | 1/111 (1)
Emotional disorder (Psychiatric disorders) | 0/120 (0) | 1/111 (1)
Euphoric mood (Psychiatric disorders) | 0/120 (0) | 1/111 (1)
Insomnia (Psychiatric disorders) | 2/120 (3) | 3/111 (5)
Libido decreased (Psychiatric disorders) | 0/120 (0) | 4/111 (4)
Mood altered (Psychiatric disorders) | 1/120 (1) | 0/111 (0)
Nightmare (Psychiatric disorders) | 0/120 (0) | 1/111 (1)
Sleep disorder (Psychiatric disorders) | 1/120 (1) | 0/111 (0)
Tearfulness (Psychiatric disorders) | 1/120 (1) | 0/111 (0)
Dysuria (Renal and urinary disorders) | 0/120 (0) | 1/111 (1)
Haematuria (Renal and urinary disorders) | 0/120 (0) | 1/111 (1)
Micturition disorder (Renal and urinary disorders) | 0/120 (0) | 1/111 (1)
Nephrolithiasis (Renal and urinary disorders) | 0/120 (0) | 1/111 (1)
Urinary hesitation (Renal and urinary disorders) | 0/120 (0) | 3/111 (3)
Urinary retention (Renal and urinary disorders) | 0/120 (0) | 1/111 (1)
Urine flow decreased (Renal and urinary disorders) | 0/120 (0) | 2/111 (2)
Ejaculation disorder (Reproductive system and breast disorders) | 0/120 (0) | 1/111 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0/120 (0) | 1/111 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 0/120 (0) | 1/111 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/120 (1) | 0/111 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/120 (0) | 1/111 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/120 (2) | 0/111 (0)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 2/120 (2) | 0/111 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/120 (1) | 1/111 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0/120 (0) | 1/111 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0/120 (0) | 1/111 (1)
Rash (Skin and subcutaneous tissue disorders) | 1/120 (1) | 1/111 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1/120 (1) | 0/111 (0)
Nail operation (Surgical and medical procedures) | 1/120 (1) | 0/111 (0)
Oral surgery (Surgical and medical procedures) | 0/120 (0) | 1/111 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1/120 (1) | 0/111 (0)
Hot flush (Vascular disorders) | 1/120 (1) | 0/111 (0)
Hypertension (Vascular disorders) | 1/120 (1) | 4/111 (4)
Hypotension (Vascular disorders) | 0/120 (0) | 1/111 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days